CLINICAL TRIAL: NCT04954534
Title: Exploratory Efficacy Study of NEUROSTEM® in Subjects Who Control Group of NEUROSTEM® Phase-I/IIa Clinical Trial
Brief Title: Exploratory Efficacy Study of NEUROSTEM® in Subjects Who Control Group of NEUROSTEM®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Principal Investigator, Duk Lyul Na, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC-CR-01
Record Dates: First submitted 2021-06-01; First posted 2021-07-08 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEUROSTEM (hUCB-MSCs) - high dose (Experimental): human umbilical cord blood-derived mesenchymal stem cells High dose: 3 x 10^7 cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4-week intervals
  Interventions: Biological: human umbilical cord blood derived mesenchymal stem cells

INTERVENTIONS:
Biological: human umbilical cord blood derived mesenchymal stem cells — High dose: 3 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4-week intervals
  Other Names: NEUROSTEM

SUMMARY:
This study is to evaluate of Exploratory Efficacy of NEUROSTEM® in Subjects who control group of NEUROSTEM® Phase-I/IIa Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have been treated with placebo in phase 1/2a clinical trial of NEUROSTEM®
2. Subjects who voluntarily decided to participate and signed the consent form after receiving explanations on the clinical trial (in case it is difficult for the participant to sign, the consent of the legal representative)

Exclusion Criteria:

1. History of stroke within 3 months prior to study enrollment
2. Severe liver disorder (equivalent to double the normal values of ALT and AST) at Visit 1
3. Severe kidney disorder (serum creatinine ≥1.5mg/dL) at Visit 1
4. Abnormal Laboratory findings at Visit 1

   * Hemoglobin < 9.5 g/dL for male and <9.0 g/dL for female
   * Total WBC Count < 3000/mm3
   * Total Bilirubin >= 3 mg/dL
5. Suspected active lung disease based on chest X-ray at Visit 1
6. Bleeding disorder (abnormal blood coagulation test result (i.e. platelet count of < 137,000/mm3, PT ≥ 1.5 INR, or aPTT ≥ 1.5 x control anti-coagulant or anti-platelet, without anticoagulant or anti-platelet therapy)
7. Diagnosis of cancer (of any body system, including brain tumor)
8. Contraindicated for any of the tests performed during the clinical trial period (for example, MRI, CT, PET)
9. Whom the principal investigator considers inappropriate for participation in the study due to any reasons other than those listed above

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-07-12 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in ADAS-Cog | 4weeks,8weeks,12weeks,24 weeks after the first dose
  The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis using an 11-point AD Assessment Scale. It has a minimum score of 0 and a maximum severity score of 70, and a higher score indicates more impairment.

SECONDARY OUTCOMES:
Change in CDR-SOB | 24 weeks after the first dose
  The CDR-SOB(Clinical Dementia Rating, Sum of Boxes) is a global rating of dementia severity based on the clinician's interpretation of the history and examination. The range of this instrument is 0 to 18 with higher numbers indicating greater impairment.
Change from the baseline in K-MMSE(korean version) | 24 weeks after the first dose
  The MMSE(Mini-Mental State Examination) is a brief, practical test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score from 0 to 30, with higher scores indicating better function
Change from the baseline in CGA-NPI | 24 weeks after the first dose
  Caregiver-administered Neuropsychiatric Inventory, Measure abnormal behavior. The score range is 0-144. A higher score means severe abnormal behavior.
Change from the baseline in SIB | 24 weeks after the first dose
  The Severe Impairment Battery (SIB) is an assessment of cognitive dysfunction across nine domains such as memory, language, and orientation. The score ranges from 0 (worst) to 100 (best)
ADAS-Cog Response Rate | The ADAS-cog response is defined as no worsening (no change or improvement on ADAS-cog score) of the ADAS-cog score at 24 weeks after the first administration compared to the baseline
  Alzheimer's Disease assessment Scale-Cognitive Subscale
Change in CIBIC-plus | 24 weeks after the first dose
  The Clinician's Interview-Based Impression of Change-plus(CIBIC-plus) is a rating scale derived from an interview with the patient and caregiver with an independent rater designed to measure several domains of patient function, such as mental/cognitive state, behavior, and activities of daily living. The scores range from 1 (marked improvement) to 7 (marked worsening).
Change from the baseline in CSF biomarkers | 24 weeks after the first dose
  biomakrers analysis (Amyloid beta 42, Phosphorylated tau, Total tau, RBC, WBC, Protein, Glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee NK, Jang H, Choi Y, Hwangbo S, Lee S, Lee JI, Kim YJ, Chin J, Chang JW, Seo SW, Son HJ, Choi SJ, Na DL, Kim HJ. Mesenchymal Stem Cells With Adjuvant Dexamethasone in Patients With Alzheimer's Disease: A Phase IIa Trial. Dement Neurocogn Disord. 2025 Oct;24(4):272-285. doi: 10.12779/dnd.2025.24.4.272. Epub 2025 Oct 24. PMID 41220869